CLINICAL TRIAL: NCT07407530
Title: Comparison of 'Sip Til Send' Regimens Prior to Elective Caesarean Delivery Using Bedside Gastric Ultrasound: a Randomized Study Comparing Water With Carbohydrate-rich Drink
Brief Title: Comparison of 'Sip Til Send' Regimens Prior to Elective Caesarean Delivery Using Bedside Gastric Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Rotunda Hospital (Other)
Responsible Party: Principal Investigator, Ryan Howle, Consultant Anaesthesiologist, The Rotunda Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: REC2025-005
Record Dates: First submitted 2025-07-17; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gastric Emptying; Caesarean Delivery; Pregnancy
Keywords: gastric ultrasound; gastric emptying; cesarean section; pregnancy; fasting guidelines

STUDY DESIGN:
Intervention Model Description: Prospective randomized single-blinded study. Randomization to intervention which will be "water" group and "carbohydrate" group.
  Pregnant women cannot be blinded to the intervention, but the healthcare workers and the investigators will be blinded to the intervention
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Sip Til Send' with water (Other): The "water" group who will be encouraged to sip at a maximum rate of 1 cup (170ml) per hour whilst waiting in hospital for an elective CD planned under neuraxial anaesthesia. The water group represent the control or standard practice group as this is in line with current hospital policy.
  Interventions: Drug: The "water group"
- 'Sip Til Send' with carbohydrate-rich drinks (Active Comparator): the "carbohydrate" group will be encouraged to sip a standardised carbohydrate-rich drink ,flavoured clear, carbohydrate drink " Nutricia preOp".
  Interventions: Drug: The carbohydrate group represent the interventional group and will utilise the standard carbohydrate-rich drink

INTERVENTIONS:
Drug: The carbohydrate group represent the interventional group and will utilise the standard carbohydrate-rich drink — the "carbohydrate" group will be encouraged to sip a standardised carbohydrate-rich drink at a maximum rate of 1 cup (170ml) per hour, whilst waiting in hospital for an elective CD planned under neuraxial anaesthesia. Prior to their CD, any remaining drink will be weighed to calculate to volume consumed (assuming a liquid density of 1mg/ml)
  Arms: 'Sip Til Send' with carbohydrate-rich drinks
Drug: The "water group" — women will be provided with a weighed jug of water which the participants may sip to comfort at a maximum rate of 1 cup (170ml) per hour
  Arms: 'Sip Til Send' with water

SUMMARY:
'Sip Til send' is a liberal drinking policy that replaces fasting before a caesarean delivery, meaning that women waiting in hospital can freely drink sips of water until they are called from the ward for their delivery. Studies has shown that 'Sip Til send' is safe and it improves the experience around surgery. Separate from this, drinking carbohydrate-rich drinks at specified time intervals before surgery is also recommended by international guidelines as part of a package of care aimed at enhancing recovery from surgery, and studies demonstrate that carbohydrate drinks significantly lower hunger sensation before caesarean delivery. The aim of this study is to combine these two interventions and compare the effects of sipping water against sipping carbohydrate drinks whilst waiting for a caesarean delivery and look at the stomach contents before delivery to ensure it is a safe practice and look at how women rate the quality of their recovery to see which practice is preferred. We will recruit women due to have an elective caesarean delivery whilst awake with a spinal anaesthetic at the Rotunda Hospital and only include those who are fully fasted on their arrival and would be candidates for the current 'Sip Til Send' policy. They will then be assigned to one of two groups, the "water" group who will be encouraged to sip water whilst waiting for surgery, and the "carbohydrate" group who will be encouraged to sip a standardised carbohydrate-rich drink instead. Using a bedside ultrasound machine, we will image the stomach and estimate the volume of liquid contents on two occasions; first, following recruitment to the study when fully fasted and before starting 'Sip Til Send', and second is immediately prior to surgery. Fluid intake will be closely monitored, and all participants will be asked to complete a short questionnaire the day after their delivery that asks them to rate aspects of their recovery. Participants and their newborns will not undergo any additional invasive testing for the study. Participants and their newborns will not undergo any additional invasive testing for the study, but consent will be sought to test women's urine for ketones (collected from the catheter bag during surgery). Medical notes will also be looked at after discharge to identify adverse outcomes such as nausea or vomiting during surgery and low blood sugar in the newborn. The study should run for approximately 3 to 6 months.

DETAILED DESCRIPTION:
This study is a prospective randomized single-blinded study. Randomisation to intervention which will be "water" group and "carbohydrate" group. Pregnant women cannot be blinded to the intervention, but the healthcare workers and the investigators will be blinded to the intervention.

This study will incorporate clinical practice protocols that are already in place at the Rotunda hospital. The enhanced recovery guidelines encourage consumption of carbohydrate drinks prior to arrival at hospital for surgery. This protocol was superseded by the introduction of 'Sip Til Send' with water with an aim to reduce fasting times after arrival at hospital, but adherence with both practices is variable.

The study intervention is the provision of water or a standard carbohydrate-rich drink which the participants may sip to comfort at a maximum rate of 1 cup (170ml) per hour whilst waiting in hospital for an elective CD planned under neuraxial anaesthesia. The water group represent the control or standard practice group as this is in line with current hospital policy. The carbohydrate group represent the interventional group and will utilise the same carbohydrate drinks available for enhanced recovery.

Eligible participants booked to undergo an elective CD will be recruited on the day of surgery by a member of the research team. Consideration will depend on the research team availability, expected fasting time of more than 1 hour and full adherence of European fasting guidelines at the time of study entry (6 hours for solids and 2 hours for liquids). Following recruitment, written consent is obtained and a 'fasting' gastric ultrasound will be performed in a standardised manner prior to randomisation. If a Perlas grade 2 antrum is encountered, this will be assumed to represent a full stomach (>1.5ml/kg) and the potential participant be removed from the study. To mitigate any further risk, they will be advised to fully fast, not be offered 'Sip Til Send' and the anaesthesiologist in charge of their clinical care will be informed. Any women in whom adequate views of the gastric antrum cannot be obtained in both positions will also be removed from the study. All other participants will then be randomized into the study.

Following group allocation, women will be provided with a weighed jug of water or carbohydrate drink, a 170ml cup and written instructions stating that they may drink continually to comfort up to 1 cup and hour and information on how to refill if required. Prior to their CD, any remaining drink will be weighed to calculate to volume consumed (assuming a liquid density of 1mg/ml) and participants will undergo a second gastric ultrasound scan immediately prior to surgery.

Normal clinical care will resume after this point with group allocation having no impact on care received. During surgery, a urine sample will be collected via the catheter bag following written consent and will be sent to the hospital laboratory to test for ketones. This result will also be available to the treating clinicians.

At around 24 hours after delivery (+/- 4 hours), women will be approached for a single follow-up visit where they will be asked to complete an obstetric-specific quality of recovery score (ObsQoR-10). Following discharge from hospital, medical notes will be interrogated for evidence of perioperative nausea, vomiting or aspiration and neonatal notes will also be interrogated for evidence of treated hypoglycaemia.

Gastric ultrasound is a safe non-invasive scan which will take about 10 minutes to complete. It involves placement of a curvilinear ultrasound probe on the upper abdomen whilst the participant is on their back and then their right-hand side. The head of the bed will be elevated to 45 degrees during the scan for comfort and to prevent aortocaval compression. A qualitative Perlas score is given based on whether clear liquid is seen in the antrum in each position. A Perlas 0 antrum has no fluid in either position, a Perlas 1 has clear fluid in the right-lateral position but not when semi-recumbent and a Perlas 2 score has identifiable clear fluid in both positions. Gastric antrum CSA will be calculated using horizontal and vertical calliper measurements inputted into a formula to calculate the area of an ellipse. These will also be used to estimate gastric volumes via the method below that has been validated in term pregnant women previously:

GV (mL) = 0.18 x right-lateral CSA (mm2) + 0.11 x semirecumbent CSA (mm2) - 62.4

ELIGIBILITY:
Inclusion Criteria:

* Planned caesarean delivery under regional anaesthesia
* Adhered to national fasting guidance of 6 hours for food and 2 hours for clear fluids
* Eligible for Sip Til Send

Exclusion Criteria:

* Planned general anaesthesia
* Emergency or urgent caesarean delivery
* Not fasted at time of recruitment
* Unable to visualise stomach or Perlas 2 stomach identified at time of recruitment
* Obesity of BMI >40
* Previous upper GI or bariatric surgery
* Age <18 years
* Insulin dependent diabetes mellitus (type 1 or 2)
* Gestational diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 190 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
24-hour Obstetric Quality of Recovery-10 (ObsQoR-10) scores | From enrollment to around 24 hours after delivery (+/- 4 hours).
  Compare the 24-hour quality of recovery scores : At around 24 hours after delivery (+/- 4 hours), women will be approached for a single follow-up visit where they will be asked to complete an obstetric-specific quality of recovery score (ObsQoR-10). This is scale from 0 to 100, with a higher number indicating a better quality of recovery.
Gastric antrum CSA | From enrollment until just before their cesarean delivery.
  Compare the gastric antrum CSA immediately prior to caesarean delivery: 'fasting' gastric ultrasound will be performed in a standardised manner prior to randomization, Prior to their CD, participants will undergo a second gastric ultrasound scan immediately prior to surgery.

SECONDARY OUTCOMES:
Estimated residual gastric volume before CD | From enrollment until just before their cesarean delivery.
  Compare the estimated residual gastric volumes prior to caesarean delivery : Gastric antrum CSA will be calculated using horizontal and vertical calliper measurements inputted into a formula to calculate the area of an ellipse. These will also be used to estimate gastric volumes via the method below that has been validated in term pregnant women previously:
  GV (mL) = 0.18 x right-lateral CSA (mm2) + 0.11 x semirecumbent CSA (mm2) - 62.4
Incidence of a full stomach assessed by quantitative ultrasound measurements | From enrollment until just before their cesarean delivery.
  Compare the incidence of estimated residual gastric volumes >1.5ml/kg
Qualitative ultrasound guided incidence of a full stomach | From enrollment until just before their cesarean delivery.
  Compare the incidence of Perlas 2 scores : A qualitative Perlas score is given based on whether clear liquid is seen in the antrum in each position. A Perlas 0 antrum has no fluid in either position, a Perlas 1 has clear fluid in the right-lateral position but not when semi-recumbent and a Perlas 2 score has identifiable clear fluid in both positions
Compare the maternal urinary ketones during caesarean delivery | From enrollment until just before their cesarean delivery.
  During surgery, a urinary catheter is inserted as part of standard clinical care. A urine sample will be collected from this prior to delivery and sent to the lab to test for ketones.
Gastric antrums CSA Vs Estimated gastric volumes | From enrollment until just before their cesarean delivery.
  Compare the average difference in gastric antrum CSA and estimated gastric volume over the course of 'Sip Til Send'
Incidence of treated neonatal hypoglycaemia | Immediately after birth
  Compare the incidence of treated hypoglycaemia in the neonates: following discharge from hospital, medical neonatal notes will be interrogated for evidence of treated hypoglycaemia

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - Rotunda Hospital, Dublin, Ireland/County Dublin
  - Rotunda Hospital, Dublin